CLINICAL TRIAL: NCT02523261
Title: Interest of Direct Aspiration First Pass Technique (ADAPT) for Thrombectomy Revascularisation of Large Vessel Occlusion in Acute Ischaemic Stroke
Acronym: ASTER
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fondation Ophtalmologique Adolphe de Rothschild (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MPN_2015_22
Record Dates: First submitted 2015-08-12; First posted 2015-08-14 (Estimated); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Ischemic Cerebrovascular Accident
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ADAPT (Experimental)
  Interventions: Procedure: direct aspiration procedure
- Stent Retriever (Active Comparator)
  Interventions: Procedure: stent retriever procedure

INTERVENTIONS:
Procedure: direct aspiration procedure — Revascularization by endovascular thrombectomy using the distal aspiration first pass technique
  Arms: ADAPT
Procedure: stent retriever procedure — Revascularization by endovascular thrombectomy using a mechanical thrombectomy device
  Arms: Stent Retriever

SUMMARY:
Mechanical thrombectomy (TM) is now validated through 4 randomized controlled trials of high scientific level as the reference treatment of cerebral infarction associated with proximal cerebral occlusion (MR CLEAN, ESCAPE 2014, 2015). These studies have shown for the first time a major decrease (-35%) of disability related to severe cerebral infarction and reduction in mortality. These studies only used thrombectomy devices called stent retriever for obtaining recanalization rates ranging from 58-72% for the 2 largest studies (MR CLEAN, ESCAPE 2014, 2015). This criterion "recanalization" is important because it largely determines the functional prognosis of patients with severe cerebral infarction (Khatri, 2014).

These results are exciting but we can do even better. Indeed, already new thrombectomy devices are available with a special interest for ADAPT (A Direct Aspiration First Pass Technic). This distal suction system, with a high level of endovascular navigability, provides high recanalization rates (> 90%), low morbidity, with a synergistic effect with stent retriever (Turk A, Kowoll 2014 and 2015). To date, these technic (ADAPT) has never been assessed in a randomized controlled trial.

We have previously conducted a comparative observational study between two recanalization strategies by thrombectomy using first-line ADAPT or the most widely used stent retriever. The interventional neuroradiologist could, in case of recanalization failure with the Solitaire system, used another thrombectomy material left to the operator's choice. 244 consecutive patients on two centers (Rothschild Foundation, and Foch Hospital, France) admitted for a cerebral infarction associated with proximal occlusion were included. This is so far the largest series of patients with ADAPT system. The complete recanalization rate was 84% with ADAPT versus 68% with stent retriever (P = 0.006). Unpublished data, Oral presentation at the European Stroke Organization, April 2015). Our research aims to show that a first line strategy of recanalization by thrombectomy using a distal suction system (ADAPT) is superior that the use of a stent retriever.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years with no upper age limit.
* Cerebral infarction in the anterior circulation
* Occlusion of the anterior circulation proven by CT angiography or MR angiography
* With or without previous Intravenous thrombolysis
* Start of thrombectomy procedure within 6 hours of symptoms onset.
* Patient expresses verbally his non-opposition to be enrolled in the study ; in case patient cannot communicate, verbal non-opposition is obtained from his close / trusted person

Exclusion Criteria:

* Absence of indication for thrombectomy
* Cons-indication for thrombectomy
* Presence of cerebral infarction of the posterior circulation
* Occlusion of the cervical carotid artery
* Allergy to x-ray contrast products
* Patient was bedridden or using a wheelchair most of the day (pre-event modified Rankin Scale score > 3) prior to stroke
* Pregnancy or breastfeeding
* Patient under legal protection
* No affiliation to health insurance

Secondary exclusion criteria

- Lack of access route for catheterization

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 381 (Actual)
Dates: Start 2015-10-10 (Actual); Primary Completion 2016-10 (Actual); Study Completion 2017-02 (Actual)

PRIMARY OUTCOMES:
Complete recanalization percentage | Immediately after the revascularization procedure is completed
  Proportion of patients in which complete recanalization is achieved as defined by a TICI score equal to 2b or 3

CONTACTS AND LOCATIONS:
Overall Officials: Michel PIOTIN, Principal Investigator — Fondation ophtalmologique de Rothschild
Locations (8):
- France (8):
  - CHU Pellegrin, Bordeaux
  - Hospices Civils de Lyon, Bron
  - CHU Dupuytren, Limoges
  - CHU Hôpital Gui de Chaulac, Montpellier
  - Hôpital Neurologique, Nancy
  - Hôpital Guillaume et René LAENNEC, Nantes
  - Fondation Ophtalmologique Adolphe de Rothschild, Paris
  - Hôpital Foch, Suresnes

REFERENCES:
- [Derived] Maier B, Robichon E, Bourcier R, Dargazanli C, Labreuche J, Thion LA, Leguen M, Riem R, Desilles JP, Boulouis G, Delvoye F, Hebert S, Redjem H, Smajda S, Escalard S, Blanc R, Piotin M, Lapergue B, Mazighi M; ASTER Trialdagger. Association of Hypotension During Thrombectomy and Outcomes Differs With the Posterior Communicating Artery Patency. Stroke. 2021 Aug;52(9):2964-2967. doi: 10.1161/STROKEAHA.121.034542. Epub 2021 Jun 17. PMID 34134507
- [Derived] Derraz I, Pou M, Labreuche J, Legrand L, Soize S, Tisserand M, Rosso C, Piotin M, Boulouis G, Oppenheim C, Naggara O, Bracard S, Clarencon F, Lapergue B, Bourcier R; ASTER and the THRACE Trials Investigators. Clot Burden Score and Collateral Status and Their Impact on Functional Outcome in Acute Ischemic Stroke. AJNR Am J Neuroradiol. 2021 Jan;42(1):42-48. doi: 10.3174/ajnr.A6865. Epub 2020 Nov 12. PMID 33184069
- [Derived] Ducroux C, Piotin M, Gory B, Labreuche J, Blanc R, Ben Maacha M, Lapergue B, Fahed R; ASTER Trial investigators. First pass effect with contact aspiration and stent retrievers in the Aspiration versus Stent Retriever (ASTER) trial. J Neurointerv Surg. 2020 Apr;12(4):386-391. doi: 10.1136/neurintsurg-2019-015215. Epub 2019 Aug 30. PMID 31471527
- [Derived] Rosso C, Blanc R, Ly J, Samson Y, Lehericy S, Gory B, Marnat G, Mazighi M, Consoli A, Labreuche J, Saleme S, Costalat V, Bracard S, Desal H, Piotin M, Lapergue B; ASTER Trial and Pitie-Salpetriere Investigators. Impact of infarct location on functional outcome following endovascular therapy for stroke. J Neurol Neurosurg Psychiatry. 2019 Mar;90(3):313-319. doi: 10.1136/jnnp-2018-318869. Epub 2018 Nov 13. PMID 30425161
- [Derived] Guenego A, Lecler A, Raymond J, Sabben C, Khoury N, Premat K, Botta D, Boisseau W, Maier B, Ciccio G, Redjem H, Smajda S, Ducroux C, Di Meglio L, Davy V, Olivot JM, Wang A, Duplantier J, Roques M, Krystal S, Koskas P, Collin A, Ben Maacha M, Hamdani M, Zuber K, Blanc R, Piotin M, Fahed R; Aspiration versus STEnt-Retriever (ASTER) trial investigators. Hemorrhagic transformation after stroke: inter- and intrarater agreement. Eur J Neurol. 2019 Mar;26(3):476-482. doi: 10.1111/ene.13859. Epub 2018 Dec 7. PMID 30414302
- [Derived] Fahed R, Ben Maacha M, Ducroux C, Khoury N, Blanc R, Piotin M, Lapergue B; ASTER Trial Investigators. Agreement between core laboratory and study investigators for imaging scores in a thrombectomy trial. J Neurointerv Surg. 2018 Dec;10(12):e30. doi: 10.1136/neurintsurg-2018-013867. Epub 2018 May 14. PMID 29760012
- [Derived] Lapergue B, Blanc R, Gory B, Labreuche J, Duhamel A, Marnat G, Saleme S, Costalat V, Bracard S, Desal H, Mazighi M, Consoli A, Piotin M; ASTER Trial Investigators. Effect of Endovascular Contact Aspiration vs Stent Retriever on Revascularization in Patients With Acute Ischemic Stroke and Large Vessel Occlusion: The ASTER Randomized Clinical Trial. JAMA. 2017 Aug 1;318(5):443-452. doi: 10.1001/jama.2017.9644. PMID 28763550
- [Derived] Blanc R, Redjem H, Ciccio G, Smajda S, Desilles JP, Orng E, Taylor G, Drumez E, Fahed R, Labreuche J, Mazighi M, Lapergue B, Piotin M. Predictors of the Aspiration Component Success of a Direct Aspiration First Pass Technique (ADAPT) for the Endovascular Treatment of Stroke Reperfusion Strategy in Anterior Circulation Acute Stroke. Stroke. 2017 Jun;48(6):1588-1593. doi: 10.1161/STROKEAHA.116.016149. Epub 2017 Apr 20. PMID 28428348